CLINICAL TRIAL: NCT05180526
Title: A Multicenter, Prospective, Post-marketing Evaluation of QLETLI (Adalimumab Injection) Treatment Clinical Study on Efficacy and Safety of Non-infectious Uveitis (UV)
Brief Title: Assessment of Safety , Clinical Efficacy with QLETLI in Non-infectious Uveitis (UV)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT-1406-006-CR
Record Dates: First submitted 2021-12-07; First posted 2022-01-06 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): 80 mg was given subcutaneously at week 1, followed by 40 mg of Glorio (adamuzumab injection) every other week from week 1 to week 22 (12 doses).
  Interventions: Drug: QLETLI

INTERVENTIONS:
Drug: QLETLI — 80 mg was given subcutaneously at week 1, followed by 40 mg of Glorio (adamuzumab injection) every other week from week 1 to week 22 (12 doses).

SUMMARY:
This is a multicenter, prospective, post-marketing clinical study with a total of 60 uveitis (UV) subjects planned to be enrolled.

Screening period (-2~0 weeks) ,Treatment period (1-22 weeks), Follow-up period, At the same time, plasma concentration will be determined

DETAILED DESCRIPTION:
This is a multicenter, prospective, post-marketing clinical study with a total of 60 uveitis (UV) subjects planned to be enrolled.

Screening period (-2~0 weeks) : the inclusion and exclusion criteria were evaluated, and those meeting the criteria could enter the treatment period.

Treatment period (1-22 weeks) : Eligible subjects with non-infectious uveitis were given an initial subcutaneous injection of 80 mg at week 1, followed by a subcutaneous injection of 40 mg of Glorio (adamuzumab injection) every other week from week 1 to week 22 (a total of 12 doses).

Follow-up period: Follow-up for safety and/or efficacy is recommended at 6, 12, 24, and 32 weeks after initiation of the study drug. A final visit will be made at 32 weeks. During the study, if the condition of the subjects or their symptoms and signs become worse, the investigator can adjust the use of drugs for uveitis other than study drugs according to the actual situation of the subjects.

At the same time, plasma concentration will be determined before D1, D78 (week 12), and D162 (week 24); Immunogenicity analysis was performed before D1 administration, before D78 (week 12), before D162 (week 24) and before D218 (week 32)

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily participated in the study and signed informed consent
* Aged between 18 and 70 (including threshold), male or female;
* Diagnosis of non-infectious intermediate, posterior, or total uveitis in at least one eye;
* Received maintenance therapy (oral prednisone 10-60mg/day or equivalent glucocorticoid for ≧2 weeks before screening, and no dose adjustment from screening to baseline;
* At baseline, at least one eye was diagnosed with active uveitis, presenting as meeting at least one of the following criteria: active inflammatory chorioretinal and/or inflammatory retinal vasculopathy; Cell grade of anterior chamber ≧2+; Degree of vitreous turbid ≧2+;
* Negative serum pregnancy test results of women of childbearing age during screening visits;

Exclusion Criteria:

* Patients with the following eye conditions:
* Patients with simple anterior uveitis;
* Uveitis with macular edema as the only manifestation;
* is confirmed or suspected infectious uveitis (including but not limited to the following causes of infectious uveitis, tuberculosis, cytomegalovirus, lyme disease, toxoplasmosis, human, T, Whipple's disease virus type 1 infection, herpes zoster virus and herpes simplex virus) or disguise syndrome (for example: eye trauma, lymphoma, malignant tumor, or surgery, etc.);
* Uncontrolled glaucoma, defined as intraocular pressure higher than 25 mmHg after drug treatment, or optic nerve damage;
* Best corrected visual acuity of less than 20 letters in at least one eye at baseline;
* With other fundus diseases (such as fertile or serious non fertile diabetic retinopathy or diabetic retinopathy with clinical significance of macular edema, retinal vein occlusion, macular degeneration, age, sex, blood vessel patterns change, the pathological myopia, retinal detachment, macular hole, toxoplasmosis, optic nerve disease, etc.);
* Demyelinating disease (including myelitis and optic neuritis) or a history of neurology suggesting symptoms of demyelinating disease (including but not limited to optic neuritis);
* Refractive media opacity or pupil failure that significantly interferes with visual acuity detection, anterior segment and fundus assessment;
* One-eyed patients deemed unsuitable for inclusion by the investigator;
* Peribulbar, intravitreal or subocular corticosteroid injections were given within 30 days prior to screening;
* Posterior capsulotomy was performed within 30 days prior to screening;
* Cataract surgery is expected within 90 days prior to screening or during the study period;
* An intravitreal injection of anti-VEGF therapy (e.g., raizumab, apecivir, or Combocept) within 90 days prior to baseline;
* Ozurdex implants (dexamethasone implants) were performed within 6 months prior to baseline;
* Treatment with intravitreal injection of methotrexate within 90 days prior to baseline;
* Had been treated with vitreous Retisert (glucocorticoid implant) or had complications with the implant during the 36 months prior to baseline; Removal of Retisert within 90 days prior to baseline or complications of removal.
* Having any of the following general conditions:
* Subjects meet any of the following criteria associated with latent or active tuberculosis (TB) infection:

  . A history of active TB ≤ 3 years before screening (but can also be included if it is > 3 years and documented completion of adequate treatment); B. Signs or symptoms suggestive of active TB at the time of screening in the history and/or physical examination; C. Recent close contact with someone with active TB; D. If a TB infection T-cell test is positive at the time of screening, subjects will be excluded from the study if their first TB infection T-cell test is inconclusive. For suitable standards has been completed before screening latent TB treatment and no other risk factors, imaging findings, or support the latent or signs of active TB specific subjects, for positive or uncertain results may be the exception handling, researchers with the qualified physician judgment, tuberculosis (including extrapulmonary) risk, decision and discuss with bidders;
* Positive hepatitis C antibody during screening; Or HIV antibody positive; Or treponema pallidum antibody positive;
* Symptoms of severe, progressive or uncontrollable kidney, liver, blood, gastrointestinal, lung, cardiovascular, neurological or brain disease. The investigator felt that participating in the study placed patients at unacceptable risk.
* Patients with malignant tumors.
* Patients with moderate to severe heart failure (New York Heart Society Grades 3-4).
* History of severe allergy or anaphylactoid reaction to monoclonal antibodies.
* Prior treatment with anti-TUMOR necrosis factor TNF or other biological agents with potential therapeutic effect for uveitis (excluding intravitreal anti-VEGF drugs).
* During the 30 days prior to baseline, the combined dose of other immunosuppressant therapy increased or did not meet any of the following conditions: methotrexate MTX≤25mg/ week; Cyclosporine ≤4 mg/kg/ day; Mycophenolate (or equivalent dose of mycophenolate) ≤2g/ day; Azathioprine ≤175 mg/ day; Tacrolimus oral ≤8 mg/ day.
* Received clinical trial drug intervention within 3 months prior to screening.
* Received any live vaccine within 3 months prior to receiving the first dose of the study drug, or planned to receive live vaccine during the study period.
* There are contraindications to dilatation drugs.
* Patients judged unsuitable for inclusion by other investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Duration of treatment failure | 6\12\24week
  Duration of treatment failure at 6 weeks of treatment or between 6 and 24 weeks of treatment (treatment failure is defined as meeting at least one of the following conditions in at least one eye:

SECONDARY OUTCOMES:
treatment failure rate | 6/12/24week
  Treatment failure rate at each visit point from first administration to 24 weeks.Treatment failure was defined as meeting at least one of the following conditions in at least one eye: newly active inflammatory choroiditis or retinal vasculopathy [from baseline]; The anterior chamber cell grading or vitreous opacity grading did not reach ≦0.5+ during the 6 weeks visit, or the optimal condition did not improve in all visits after 6 weeks. Best corrected visual acuity decreased by ≧15 letters compared to best condition
Changes in ocular inflammation | 6/12/24week
  changes in anterior chamber cell grade
Changes in ocular inflammation | 6/12/24week
  changes in vitreous turbidity
Changes in ocular inflammation | 6/12/24week
  changes in macular edema
Changes in ocular inflammation | 6/12/24week
  changes in central retinal thickness
Changes in visual acuity | 6/12/24week
  Changes in visual acuity
Changes in visual function scale VFQ-25 | 6/12/24week
  Changes in visual function scale VFQ-25

CONTACTS AND LOCATIONS:
Overall Officials: Peizeng Yang, M.D, Principal Investigator — 1 Youyi Road, Yuzhong District, Chongqing, China
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The second hospital of Jilin University, Jilin
  - Tianjin Medical University Eye Hospital, Tianjin
  - Renmin Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No